CLINICAL TRIAL: NCT07218692
Title: A Phase 2 Study of RP2 With Tivozanib in Patients With Metastatic Renal Carcinoma After Progression to Immunotherapy
Brief Title: RP2 and Tivozanib for the Treatment of Metastatic Renal Cell Cancer After Progression on Immunotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25317; NCI-2025-07332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25317 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Advanced Renal Cell Carcinoma; Advanced Sarcomatoid Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Sarcomatoid Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — Biopsy; Specimen Handling; tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (RP2, tivozanib) (Experimental): Patients receive RP2 intratumorally on days 1, 15, 29, 43, 64, 85, 106, and 127. Treatment repeats every 2 weeks for the first 4 doses and then every 3 weeks for subsequent doses for up to 8 doses in the absence of disease progression or unacceptable toxicity. After completion of the first course of treatment, patients who meet criteria may receive another course of RP2 intratumorally every 3 weeks for up to an additional 8 doses. Patients also receive tivozanib PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT and urine and blood sample collection throughout the study. Additionally, patients may undergo tumor biopsies throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Sturlimogene Erparepvec; Drug: Tivozanib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Sturlimogene Erparepvec — Given intratumorally
  Other Names: Oncolytic Herpes Simplex Virus-1 Expressing Anti-CTLA-4 Antibody-like Molecule and GM-CSF RP2; Oncolytic Herpes Simplex Virus-1 Expressing Anti-CTLA-4 Antibody-like Molecule/GM-CSF RP2; Oncolytic HSV-1 Expressing Anti-CTLA-4 Antibody-like Molecule and GM-CSF RP2; Oncolytic HSV-1 Expressing Anti-CTLA-4 Antibody-like Molecule/GM-CSF RP2; Oncolytic Virus RP2; RP 2; RP-2; RP2
Drug: Tivozanib — Given PO
  Other Names: AV 951; AV-951; AV951

SUMMARY:
This phase II trial tests the effect of RP2 and tivozanib in treating patients with renal cell cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and that is growing, spreading, or getting worse (progressive) after receiving immunotherapy with immune checkpoint inhibitors (ICIs). RP2 is a herpes simplex virus (a viral infection commonly known as the "cold sore virus") that has been changed to infect and destroy tumor cells and to activate (turn on) the human immune system to attack the tumor cells. Tivozanib hydrochloride blocks certain proteins, which may help keep tumor cells from growing. It may also prevent the growth of new blood vessels that tumors need to grow. Tivozanib hydrochloride is a type of tyrosine kinase inhibitor and a type of antiangiogenesis agent. Giving RP2 and tivozanib may be safe, tolerable, and/or effective in treating patients with metastatic renal cell cancer that has progressed after receiving immunotherapy with ICIs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the overall response rate (ORR) of the combination of sturlimogene erparepvec (RP2) with tivozanib in patients with metastatic clear cell renal carcinoma after immediate progression to first-line immunotherapy with an anti-PD1 antibody.

SECONDARY OBJECTIVES:

I. To characterize the safety and toxicity associated with the combination therapy of RP2 with tivozanib in patients with metastatic clear cell renal carcinoma after immediate progression to first-line immunotherapy with an anti-PD1 antibody.

II. To characterize the population of patients that receive RP2 with tivozanib as a subsequent line treatment.

III. To determine the progression-free survival (PFS) associated with the combination therapy of RP2 with tivozanib in patients with metastatic clear cell renal carcinoma after immediate progression to first-line immunotherapy with an anti-PD1 antibody.

IV. To determine the overall survival (OS) associated with the combination therapy of RP2 with tivozanib in patients with metastatic clear cell renal carcinoma after immediate progression to first-line immunotherapy with an anti-PD1 antibody.

OUTLINE:

Patients receive RP2 intratumorally on days 1, 15, 29, 43, 64, 85, 106, and 127. Treatment repeats every 2 weeks for the first 4 doses and then every 3 weeks for subsequent doses for up to 8 doses in the absence of disease progression or unacceptable toxicity. After completion of the first course of treatment, patients who meet criteria may receive another course of RP2 intratumorally every 3 weeks for up to an additional 8 doses. Patients also receive tivozanib orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) and urine and blood sample collection throughout the study. Additionally, patients may undergo tumor biopsies throughout the study.

After completion of study treatment, patients are followed up at 30 days then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Must be willing to consent to provide fresh tumor biopsy sample or archival tumor biopsy sample obtained within 90 days before the first dose of study treatment

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Male or female who is 18 years of age or older at the time of signed informed consent
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Histologically confirmed renal cell carcinoma with a clear-cell or sarcomatoid component
* Patients must have received exactly one prior line or two prior lines of systemic therapy in the advanced or metastatic setting, including mandatory exposure to both an immune checkpoint inhibitor (ICI) and one antiangiogenic tyrosine kinase inhibitor (TKI). Prior treatment with hypoxia inducible factor (HIF)-α inhibitors is not permitted. Patients who received adjuvant immunotherapy and experienced disease recurrence within 6 months of completing treatment may also be eligible, and such therapy will count toward prior lines
* Has injectable tumor(s), which alone or in aggregate, total at least 1 cm in diameter of RP2
* Has at least 1 measurable tumor of ≥ 1 cm in longest diameter (or ≥ 1.5 cm shortest diameter for lymph nodes) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* White blood cell (WBC) count ≥ 2.0 x 10^9/L
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets ≥ 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin ≥ 9g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN
* Creatinine clearance of ≥ 30 mL/min per the Cockcroft-Gault formula or serum creatinine < 1.5 x upper limit of normal (ULN)
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* Left ventricular ejection fraction (LVEF) ≥ 50%

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* QT interval corrected for heart rate using Bazetts's formula (QTcB) ≤ 480 ms

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP) must have a negative serum beta-human chorionic gonadotropin (β-hCG) test with a minimum sensitivity of 25 IU/L or equivalent units of β-hCG within 72 hours before the first dose and a negative urine pregnancy test on dose 1 day 1
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at and for at least (a) 90 days after the last dose of RP2 or for one month after the last dose of tivozanib. Men must also agree to refrain from donating sperm during the treatment period and for at least 90 days after the last dose of RP2

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Received a live vaccine within 28 days before the first dose of study treatment

  * Note: Seasonal influenza vaccines for injection or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines are generally inactivated vaccines and are allowed. Live/attenuated vaccines (such as the intranasal influenza vaccines) are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study treatment

  * Note: Patients who have entered the follow-up phase of an investigational study may participate if it has been 4 weeks after the last dose of the previous investigational agent
* Systemic anticancer therapies within 4 weeks of the first dose of study drug. The prior anti-PD-1 or anti-PD-L1 containing regimen is excluded from this requirement
* Received prior treatment with an oncolytic virus therapy
* Received radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities (except for radiation-induced xerostomia), not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease

  * Note: Patients must have recovered (to grade ≤ 1 or baseline) from all adverse events (AEs) due to previous therapies. Patients with grade ≤ 2 neuropathy may be eligible if approved by the medical monitor
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* History of allergy or sensitivity to study drug components or prior monoclonal antibody treatment; known hypersensitivity to Chinese hamster ovary cell products
* Known human immunodeficiency virus (HIV) infection
* Known acute or chronic hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known acute or chronic hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected)

  * Note 1: If HCV RNA testing not available, may use quantitative HCV RNA testing (preferred) or qualitative HCV antibody detection
  * Note 2: For patients with known acute or chronic hepatitis B virus (HBV) and/or HCV infection, HBV and/or HCV viral load by real-time polymerase chain reaction (qPCR) must be below the limit of quantitation for the laboratory test used, and they must not have had recent treatment within 12 weeks for HBV or HCV with antiviral medications. Patients with acute or chronic HBV or HCV must be expected to not require antiviral therapy during the RP2 treatment period
* Clinically significant uncontrolled illness
* Active significant herpetic infections or prior complications of herpes simplex virus 1 (HSV-1) infection (eg, herpetic keratitis or encephalitis) or requires intermittent or chronic use of systemic (oral or intravenous [IV]) antivirals with known antiherpetic activity (eg, acyclovir)

  * Note: Patients with sporadic cold sores may be enrolled if no active cold sores are present at the time of dose 1 day 1
* Systemic infection requiring IV antibiotics or other serious infection within 14 days before dosing
* Significant bleeding event within the last 12 months that places the patient at unjustifiable risk for bleeding from intratumoral injection procedures, based on Investigator or interventional radiologist assessment
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis
* History of interstitial lung disease, idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), non-infectious pneumonitis that required steroids, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

  * Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active tuberculosis
* History or evidence of psychiatric, substance abuse, or any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the investigator or the medical monitor, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion
* Active, known, or suspected autoimmune disease requiring systemic treatment

  * Note: Patients with type 1 diabetes mellitus and/or hypothyroidism requiring only hormone replacement, and/or with autoimmune skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, and/or prior non-serious autoimmune conditions not expected to recur are permitted to enroll
* Conditions requiring treatment with immunosuppressive doses (> 10 mg per day of prednisone or equivalent) of systemic corticosteroids within 14 days before dose 1 day 1

  * Note: Patients who require a brief course (≤ 7 days) of corticosteroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded. Physiologic replacement doses of systemic corticosteroids are permitted, only if the dose does not exceed 10 mg/day prednisone equivalent
* History of life-threatening toxicity related to prior immune therapy (eg, anti-cytotoxic T lymphocyte antigen 4 or anti-PD-1/anti-PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways [eg, CD40,4-1BB]) except those that are unlikely to recur or are expected to be manageable with standard countermeasures (eg, hormone replacement after adrenal crisis). Individual cases should be discussed with medical monitor if needed
* Conditions in which anticoagulant therapies cannot be safely stopped in the periprocedural period or patients on coumadin with a target INR > 2.5 or that cannot be temporarily reversed to INR ≤ 1.7
* Treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks before treatment
* Prior organ transplantation including allogeneic stem-cell transplantation
* Major surgery within 28 days before starting treatment or anticipated major surgery while on study

  * Note: If a patient received major surgery, they must have recovered adequately from the intervention before starting study treatment and must have adequate wound healing, based on investigator's assessment or surgeon's assessment, before starting tivozanib
* Females only: Pregnant or breastfeeding
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-08-11 (Estimated); Primary Completion 2027-08-11 (Estimated); Study Completion 2027-08-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  Will be defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) per the Response Evaluation Criteria in Solid Tumors version (v) 1.1. Will be calculated as the number of patients with CR or PR divided by the total number of treated and evaluable subjects. Will be summarized with 80% confidence intervals.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From start of treatment to progression or death, whichever occurs first, assessed up to 2 years
  Will be analyzed using Kaplan-Meier survival methods. Median PFS and corresponding 80% confidence intervals will be reported. Cox proportional hazards modeling may be used to estimate hazard ratios and corresponding confidence intervals, though formal comparisons are not powered. Results will be interpreted in an exploratory context.
Overall survival (OS) | From start of treatment to death from any cause, assessed up to 2 years
  Will be analyzed using Kaplan-Meier methods. Median OS and associated 80% confidence intervals will be reported. Cox proportional hazards modeling may be used to estimate hazard ratios. Findings will be considered descriptive and interpreted cautiously due to the single-arm nature of the trial.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs including grade 3 or greater AEs, serious AEs, and treatment-related AEs , immune-related AEs (irAEs), and AEs leading to treatment discontinuation will be assessed per Common Terminology Criteria for Adverse Events v 5.0. Will be summarized using descriptive statistics. Time to onset and resolution of irAEs will also be explored when applicable.
Baseline characteristics | At baseline
  Descriptive statistics and graphical summaries will be used to characterize the baseline demographic and clinical features of the study population, including measures of central tendency (mean, median) and frequency distributions for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Nguyen, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California